CLINICAL TRIAL: NCT04742283
Title: A Phase IIb, Randomized, Double-Masked, Active-Controlled, Parallel-Group, Multicenter Study Assessing the Efficacy and Safety of DE-126 Ophthalmic Solution 0.002% Compared With Timolol Maleate Ophthalmic Solution 0.5% in Subjects With Primary Open Angle Glaucoma or Ocular Hypertension
Brief Title: Multicenter Study Assessing the Efficacy and Safety of DE-126 Ophthalmic Solution 0.002% Compared With Timolol Maleate Ophthalmic Solution 0.5% in Subjects With Primary Open Angle Glaucoma or Ocular Hypertension
Acronym: ANGEL-2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Santen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 012604IN
Record Dates: First submitted 2021-01-28; First posted 2021-02-08 (Actual); Results first posted 2023-01-26 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Primary Open Angle Glaucoma; Ocular Hypertension
Keywords: Glaucoma
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension; Glaucoma | interventions — BID protein, human

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- DE-126 Opthalmic Solution 0.002% QD and Vehicle QD (Experimental): DE-126 Ophthalmic Solution 0.002% is administered once daily (QD)
  Interventions: Drug: DE-126 Ophthalmic Solution 0.002% QD
- Timolol Maleate Opthalmic Solution 0.5% BID (Active Comparator): Timolol Maleate Ophthalmic Solution 0.5% is administered twice daily (BID)
  Interventions: Drug: Timolol Maleate Ophthalmic Solution 0.5% BID

INTERVENTIONS:
Drug: DE-126 Ophthalmic Solution 0.002% QD — DE-126 Ophthalmic Solution QD evening and Vehicle QD Morning
  Arms: DE-126 Opthalmic Solution 0.002% QD and Vehicle QD
Drug: Timolol Maleate Ophthalmic Solution 0.5% BID — Timolol Maleate Ophthalmic Solution BID (morning and evening)
  Arms: Timolol Maleate Opthalmic Solution 0.5% BID

SUMMARY:
Reduction of elevated pressure in the eye (Intraocular pressure, or 'IOP') with eye drop medications has been shown to be effective in delaying or preventing the progression of glaucoma, and it is the only proven method for reducing the risk of glaucomatous visual field loss.

This study is being conducted to determine how well DE-126 ophthalmic solution works (efficacy) in safely lowering IOP when dosed as topical eyedrops. This study will evaluate the safety and efficacy of DE-126, ophthalmic solution in subjects with Primary Open Angle Glaucoma (POAG) or Ocular Hypertension (OHT).

The IOP will be measured at 3 different times throughout the day, over 4 total visits during a 3-month treatment period (with up to 4 extra weeks observation if the patient must stop taking current eye drops to lower IOP). Safety assessments will be done throughout the study, including ocular signs and symptoms, and vital signs. While the most important time-point to measure IOP in this study and evaluate efficacy will be at the final study visit (month 3), IOP values will also be evaluated at other visits throughout the 3-month treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Have been diagnosed of POAG or OHT in both eyes, or one eye with OAG and other with OHT
* Completed the required wait/washout period
* Qualifying Day 1 IOP measurement at 3 time-points in both eyes

Exclusion Criteria:

* Females who are pregnant, nursing, or planning a pregnancy
* Subjects who cannot safely discontinue use of ocular hypotensive medications during the wait/washout period.
* History of ocular surgery specifically intended to lower IOP in either eye. Laser iridotomy in history is allowed
* Presence of advanced glaucoma in either eye

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 323 (Actual)
Dates: Start 2020-12-17 (Actual); Primary Completion 2021-12-07 (Actual); Study Completion 2021-12-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (41):
- United States (41):
  - Arizona Eye Center, Chandler, Arizona
  - Arizona Glaucoma Specialists, Phoenix, Arizona
  - Walman Eye Center, Sun City, Arizona
  - Global Research Management, Glendale, California
  - Premiere Practice Management, Los Angeles, California
  - North Valley Eye Medical Group, Mission Hills, California
  - The Eye Research Foundation, Newport Beach, California
  - University of California, Los Angeles, Doheny Eye Centers, Pasadena, California
  - North Bay Eye Associates, Inc, Petaluma, California
  - Sacramento Eye Consultants, Sacramento, California
  - University of Colorado, Dept. of Opthamology, Aurora, Colorado
  - Hernando Eye Institute, Brooksville, Florida
  - Eye Associates of Fort Myers, Fort Myers, Florida
  - Levenson Eye Associates, Jacksonville, Florida
  - Mayo Clinic, Dept. of Opthamology, Jacksonville, Florida
  - Bowden Eye & Associates, Jacksonville, Florida
  - Shettle Eye Research, Largo, Florida
  - Dixophthal PC dba Dixon Eye Care, Albany, Georgia
  - Clayton Eye Clinical Research, LLC, Morrow, Georgia
  - Coastal Research Associates, Roswell, Georgia
  - Clinical Eye Research of Boston, LLC, Winchester, Massachusetts
  - Nevada Eye Care Professionals, Las Vegas, Nevada
  - AdvanceMed Clinical Research-Las Vegas, Las Vegas, Nevada
  - Northern New Jersey Eye Institute, South Orange, New Jersey
  - Rochester Ophthalmological Group, P.C., Rochester, New York
  - Duke Eye Center, Durham, North Carolina
  - Wake Forest Health Network Ophthamology - Oak Hollow, High Point, North Carolina
  - Vance Thompson Vision - ND, West Fargo, North Dakota
  - Apex Eye Clinical Research, LLC, Cincinnati, Ohio
  - Office of Mark J. Weiss MD, Tulsa, Oklahoma
  - Scott & Christie and Associates PC, Cranberry Township, Pennsylvania
  - Wills Eye Hospital, Philadelphia, Pennsylvania
  - Black Hills Regional Eye Institute, Rapid City, South Dakota
  - University Eye Specialists, Maryville, Tennessee
  - VRF Eye Specialty Group, Memphis, Tennessee
  - Glaucoma Associates of Texas, Dallas, Texas
  - The Cataract and Glaucoma Center, El Paso, Texas
  - DCT- Shah Research LLC dba Discovery Clinical Trials, Mission, Texas
  - San Antonio Eye Center, San Antonio, Texas
  - R and R Eye Research LLC, San Antonio, Texas
  - Stacy R. Smith M.D. P.C., Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Timolol Maleate Opthalmic Solution 0.5% BID | DE-126 Opthalmic Solution 0.002% QD and Vehicle QD
Started | 161 | 162
Completed | 148 | 158
Not Completed | 13 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Timolol Maleate Opthalmic Solution 0.5% BID | DE-126 Opthalmic Solution 0.002% QD and Vehicle QD | Total
Number analyzed (Participants) | 161 | 162 | 323
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.5 (11.63) | 66.2 (10.24) | 65.9 (10.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 83 | 86 | 169
  Male | 78 | 76 | 154
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 116 | 120 | 236
  Black or African American | 43 | 36 | 79
  Asian | 1 | 4 | 5
  American Indian or Alaska Native | 0 | 1 | 1
  Multiple | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Intraocular Pressure at Week 2
Description: Intraocular pressure (IOP), the fluid pressure inside the eye was measure by the Goldmann applanation tonometer in millimeters mercury (mmHg) at 3 time-points throughout the day. Analysis using Mixed-effects Model for Repeated Measures (MMRM).
Time Frame: 08:00, 10:00 and 16:00 at Week 2
Population: The Full Analysis Set (FAS) includes all randomized subjects who received at least one dose of the study medication (test or control medication) and had at least one post-baseline efficacy assessment of the study eye during the study.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Timolol Maleate Opthalmic Solution 0.5% BID | DE-126 Opthalmic Solution 0.002% QD and Vehicle QD
Number analyzed (Participants) | 159 | 161
mmHg
  8:00 | 19.05 (0.242) | 18.92 (0.239)
  10:00 | 18.28 (0.219) | 17.86 (0.216)
  16:00 | 17.91 (0.215) | 17.15 (0.212)

2. Primary Outcome: Intraocular Pressure at Week 6
Description: as for outcome 1
Time Frame: 08:00, 10:00 and 16:00 at Week 6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Timolol Maleate Opthalmic Solution 0.5% BID | DE-126 Opthalmic Solution 0.002% QD and Vehicle QD
Number analyzed (Participants) | 159 | 161
mmHg
  8:00 | 18.72 (0.238) | 18.32 (0.233)
  10:00 | 18.29 (0.238) | 17.96 (0.233)
  16:00 | 18.24 (0.235) | 17.52 (0.229)

3. Primary Outcome: Intraocular Pressure at Month 3
Description: as for outcome 1
Time Frame: 08:00, 10:00 and 16:00 at Month 3
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Timolol Maleate Opthalmic Solution 0.5% BID | DE-126 Opthalmic Solution 0.002% QD and Vehicle QD
Number analyzed (Participants) | 159 | 161
mmHg
  8:00 | 18.78 (0.249) | 18.80 (0.244)
  10:00 | 18.12 (0.244) | 18.07 (0.239)
  16:00 | 18.52 (0.228) | 17.57 (0.223)

4. Secondary Outcome: Mean Diurnal Intraocular Pressure at Month 3
Description: Mean diurnal Intraocular Pressure (IOP) was defined as the mean of the IOP valued at the three schedules timepoints (8:00, 10:00 and 16:00) at that visit for that subject.
Time Frame: Three months
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | Timolol Maleate Opthalmic Solution 0.5% BID | DE-126 Opthalmic Solution 0.002% QD and Vehicle QD
Number analyzed (Participants) | 159 | 161
mmHg | 18.43 (0.209) | 18.15 (0.205)

ADVERSE EVENTS:
Time Frame: From informed consent to until subject withdrawal or study exit at month 3 including two weeks of follow up after last study drug administration.
Description: Treatment emergent adverse events were summarized for the safety population. The Safety population will include all randomized subjects who received at least one dose of the study medication.
Arm/Group | Timolol Maleate Opthalmic Solution 0.5% BID | DE-126 Opthalmic Solution 0.002% QD and Vehicle QD
All-Cause Mortality (participants affected / at risk) | 0/160 | 0/161
Serious Adverse Events (participants affected / at risk) | 3/160 | 1/161
Other Adverse Events (participants affected / at risk) | 34/160 | 38/161
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Timolol Maleate Opthalmic Solution 0.5% BID (N=160) | DE-126 Opthalmic Solution 0.002% QD and Vehicle QD (N=161)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Rib Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Sternal Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Timolol Maleate Opthalmic Solution 0.5% BID (N=160) | DE-126 Opthalmic Solution 0.002% QD and Vehicle QD (N=161)
Conjunctival hyperaemia (Eye disorders) | 4 | 16
Eye pruritus (Eye disorders) | 1 | 4
Eye pain (Eye disorders) | 1 | 3
Dry eye (Eye disorders) | 2 | 2
Foreign body sensation in eyes (Eye disorders) | 1 | 2
Ocular hyperaemia (Eye disorders) | 1 | 2
Chalazion (Eye disorders) | 1 | 1
Conjunctival haemorrhage (Eye disorders) | 1 | 1
Eye irritation (Eye disorders) | 1 | 1
Eyelash thickening (Eye disorders) | 0 | 1
Eyelid margin crusting (Eye disorders) | 0 | 1
Scintillating scotoma (Eye disorders) | 0 | 1
Anterior chamber cell (Eye disorders) | 1 | 0
Anterior chamber flare (Eye disorders) | 1 | 0
Lacrimation increased (Eye disorders) | 1 | 0
Macular fibrosis (Eye disorders) | 1 | 0
Vision blurred (Eye disorders) | 1 | 0
Fatigue (General disorders) | 0 | 1
Instillation site pain (General disorders) | 6 | 1
Instillation site pruritus (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Asthenia (General disorders) | 1 | 0
Drug intolerance (General disorders) | 1 | 0
Bronchitis (Infections and infestations) | 0 | 2
COVID-19 (Infections and infestations) | 1 | 0
Onychomycosis (Infections and infestations) | 1 | 0
Tooth infection (Infections and infestations) | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1
Limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0
Blood cholesterol increased (Investigations) | 0 | 1
Vital dye staining cornea present (Investigations) | 2 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Lower respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Food allergy (Immune system disorders) | 0 | 1
Seasonal allergy (Immune system disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 1 | 0
Headache (Nervous system disorders) | 2 | 1
Depression (Psychiatric disorders) | 1 | 0
Breast mass (Reproductive system and breast disorders) | 1 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0
Madarosis (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-02-18): https://cdn.clinicaltrials.gov/large-docs/83/NCT04742283/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-15): https://cdn.clinicaltrials.gov/large-docs/83/NCT04742283/SAP_001.pdf